CLINICAL TRIAL: NCT06869148
Title: Evaluation of Prioritized Assessment for Older Patients Living With Frailty Presenting to the Emergency Department
Status: Completed | Type: Observational
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Daniel Wilhelms, Principal Investigator Daniel Wilhelms , PhD, MD . Department of Emergency Medicine in Linköping, and Department of Biomedical and Clinical Sciences, Linköping University, Linköping, Sweden, University Hospital, Linkoeping
Other Study IDs: 2024-05740-01
Record Dates: First submitted 2025-03-03; First posted 2025-03-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-03

CONDITIONS: Frailty; Length of Stay; Emergency Department Visit; Older Patients
Keywords: Clinical frailty scale; CFS; Frailty assessment; Triage; Emergency department; Length of stay; physician prioritization; physician prioritisation
MeSH Terms: conditions — Frailty; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: Patients aged 65 years or older visisting the ED who have been assessed for frailty. The control group were included before implementation of the local guidelines.
- Intervention group: Patients aged 65 years or older visisting the ED who have been assessed for frailty. The intervention group were included after the implementation of the local guidelines.
  Interventions: Other: Prioritized assessment for older patients living with frailty

INTERVENTIONS:
Other: Prioritized assessment for older patients living with frailty — In the beginning of 2025, the Emergency department of University hospital of Linköping launched a clinical guideline which stated that patients aged 65 years or older should be assessed with CFS as early as possible, preferably in connection to triage. If the patients were assessed as living with frailty, the frailty score should be stated in the electronical overview of ED patients. The patient's needs of care should be met according to frailty level and the responsible clinical team should aim to decrease the ED length of stay for older patients living with frailty.
  Other Names: Local guidelines regarding frailty in the Emergency Department
  Groups: Intervention group

SUMMARY:
The older population is getting older and growing in size worldwide. This requires healthcare to adapt to meet the complex medical and nursing needs of the older patient group. As older patients have varying health conditions with different levels of functions, their premise to handle acute, unexpected illness differs as well. This complicates matters for healthcare, especially emergency departments (ED) where resource allocation and identifying patients that are at greatest risk of negative health outcomes must be prioritized in a limited time.

When patients present to the ED, initial triage information such as vital signs and reason for visit determines the triage acuity for the patient. In Linköping, and large parts of Sweden, the triage tool RETTS (Rapid Emergency Triage and Treatment System) is used, where the highest priority is red (priority 1), then orange (priority 2), yellow (priority 3), green (priority 4) and blue (priority 5). However, this can be misleading when assessing older patients due to altered physiology with natural ageing and older patients are known to be under-triaged with existing triage systems.

The variation in functional capacity in older patients does not necessarily correlate with comorbidities and age and has been condensed to the term 'frailty'. It has been proposed that the frailty level corresponds more to biological age rather than chronological age. Frailty increases the risk of adverse outcomes such as falls, the need of in-hospital care, institutionalization, and mortality in which the risk is increased even in low acuity illnesses.

Frailty can be assessed by various means and based on the theory of cumulative deficit, frailty assessment instruments have been developed where frailty level increases with the amount of help needed from others. Different instruments have been compared in the ED and the Clinical Frailty Scale (CFS) have been deemed fit due to it being practical in a busy environment. The scale consists of 9 points where 9 is the highest level of frailty and the scale is usually dichotomized into "robust" and "living with frailty" where 5 points or above constitutes frailty. The prognostic value of CFS has previously been studied in the ED of University hospital of Linköping in Sweden with results indicating that the instrument should be used as an additional risk assessment in the ED.

Older patients often present with vague and complex symptoms to th ED, which could lead to prolonged ED stay due to the need of extensive medical workup or therapy. Long ED stays have been shown to increase both morbidity and mortality in older patients as well as risk of delirium and complications relating to care, especially in individuals living with frailty. In order to decrease the adverse events, aim to shorten ED length of stay (ED LOS) should therefore be a reasonable goal in clinical improvement work. Early identification of frailty in the ED may lead to rapid assessments and streaming of care for older patients which have shown to statistically significantly decrease ED LOS, which is why an early assessment by a physician potentially could decrease overall ED LOS. However, it is unknown how early assessed frailty could affect the ED visit itself.

In the beginning of 2025, the Emergency department of University hospital of Linköping launched a local guideline which recommended that patients aged 65 years or older visiting the ED should be assessed with CFS as early as possible, preferably in connection to triage. If the patients were assessed as living with frailty, the frailty score should be stated in the electronical overview of ED patients. The patient's needs of care should be induvidualized according to frailty level and the responsible clinical team should aim to decrease the ED length of stay for older patients living with frailty.

This study focuses on the outcomes of this newly implemented routine and aims to answer if recommended prioritization of older ED patients living with frailty leads to decreased ED LOS. Furthermore the study investigates if the clinical guidelines have an impact on time to the first assessment by a physician, admission rate, in-hospital length of stay, and mortality at 90 days

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* Assessed by CFS with the score being documented in the electronic journal

Exclusion Criteria:

* Under the age of 65 years of age
* Not assessed by CFS
* Refusal of participation in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients visiting the ED in Linköping in the age of 65 years or older who have been assessed by CFS
Sampling Method: Non-Probability Sample
Enrollment: 1217 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
ED length of stay | From enrollment until end of inclusion, approximately 4-8 weeks for each group
  Length of stay in the ED measured in hours and minutes (data will be collected from the electronic health record)

SECONDARY OUTCOMES:
Time to the first assessment by a physician | From enrollment until end of inclusion, approximately 4 weeks for each group
  Time to the first assessment by a physician (measured in minutes)
Admission rate | From enrollment until end of inclusion, approximately 4-8 weeks for each group
  Proportion of patients in each group that were admitted, measured in amount of patients and percentage.
In-hospital length of stay | From enrollment until end of inclusion, approximately 4-8 weeks for each group
  Length of in-hospital stay, measured in days.
Mortality up to 90 days | From enrollment until end of inclusion, approximately 4-8 weeks for each group
  Proportion of patients who deceased up to 90 days post ED-visit, including mortality at ED and in-hospital mortality. Measured in amount of patients and percentage.
Difference in ED length of stay between patients in different triage categories | From enrollment until end of inclusion, approximately 4-8 weeks for each group
  Difference in ED length of stay between patients in different triage categories, measured in hours and minutes. The triage categories are: Red (priority 1), orange (priority 2), yellow (priority 3), green (priority 4), and blue (priority 5).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Emergency Medicine, University hospital, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wretborn J, Munir-Ehrlington S, Horlin E, Wilhelms DB. Addition of the clinical frailty scale to triage tools and early warning scores improves mortality prognostication at 30 days: A prospective observational multicenter study. J Am Coll Emerg Physicians Open. 2024 Sep 9;5(5):e13244. doi: 10.1002/emp2.13244. eCollection 2024 Oct. PMID 39253302
- [Background] Munir Ehrlington S, Horlin E, Toll John R, Wretborn J, Wilhelms D. Frailty is associated with 30-day mortality: a multicentre study of Swedish emergency departments. Emerg Med J. 2024 Aug 21;41(9):514-519. doi: 10.1136/emermed-2023-213444. PMID 39053972
- [Derived] Ehrlington SM, Wretborn J, Wilhelms D. Frailty Alerts Reduce Waiting Time and Length of Stay in the Emergency Department. Acad Emerg Med. 2026 Feb;33(2):e70239. doi: 10.1111/acem.70239. PMID 41645916